CLINICAL TRIAL: NCT04972045
Title: Bioavailability of Curcumin Capsules in Healthy Adult Subjects: an Open, Randomized, Single-dose, Two-period, Two-sequence Crossover Study
Brief Title: Bioavailability of Curcumin Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Chenland Nutritionals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HT-PK-2021-01
Record Dates: First submitted 2021-04-05; First posted 2021-07-22 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Subjects will be given test preparation (A) or control preparation (B) on the first day of the first cycle. After a 7-day washout period, on the 8th day of the second cycle, subjects will be cross-administered with the control preparation (B) or test preparation (A)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CuminUP60®,then Curcumin capsules (Experimental): Participants first received CuminUP60® 1600mg on the first day in a fasting state.After a washout period of 7days,they then received curcumin capsules 1600mg on the eighth day in a fasting state.
  Interventions: Drug: CuminUP60®; Drug: Curcumin capsules
- Curcumin capsules,then CuminUP60® (Experimental): Participants first received curcumin capsules 1600mg on the first day in a fasting state.After a washout period of 7days,they then received CuminUP60® 1600mg on the eighth day in a fasting state.
  Interventions: Drug: CuminUP60®; Drug: Curcumin capsules

INTERVENTIONS:
Drug: CuminUP60® — 4 capsules, 400 mg / capsule
Drug: Curcumin capsules — 4 capsules, 400 mg / capsule

SUMMARY:
A single-center, open-label, randomized, two-period, crossover study design of pharmacokinetics and bioavailability in healthy adult male and female subjects under fasting conditions.

DETAILED DESCRIPTION:
Upgraded curcumin capsules(CuminUP60®) is made from curcumin with a natural extraction content of 95% and excipients through physical process microprocessing, with a curcumin content of more than 60%. CuminUP60® capsules are 400 mg/ capsules and ordinary curcumin capsules are 400 mg/ capsules. The main purpose of this study is to evaluate the bioavailability by comparing the pharmacokinetics of CuminUP60® capsule with that of curcumin capsule before the prescription improvement.

12 cases are planned to be enrolled.According to the random table, each subject will be randomly assigned to one of two groups (group 1: A/B, group 2: B/A). The cleaning period between the two doses is 7 days. Subjects were given the test preparation (A) or the control preparation (B) on the first day of the first cycle of the trial, and were temporarily allowed to leave the phase I clinical research center after 72 hours of blood sample collection and vital signs examination after the completion of the medication. After a 7-day wash period, on the 8th day of the second cycle, the subject will be cross-administered with the control formulation (B) or the test formulation (A), all procedures are the same as in the first cycle.

On the 11th day (the second cycle), subjects will undergo physical examination, ECG examination, assessment of vital signs (blood pressure, pulse, body temperature), laboratory examinations (blood biochemistry, blood routine, urine routine, detailed examination items are shown in the appendix 1) Female subjects must undergo a blood pregnancy test and then be allowed to leave the research center.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical trial, understand and voluntarily signed a written informed consent;
* Able to complete the research in accordance with the requirements of the test plan;
* Subjects (including male subjects) have taken effective contraceptive measures within 14 days before screening and are willing to have no pregnancy plan within 3 months after the end of the study and voluntarily take effective contraceptive measures;
* Male and female subjects aged 18 to 55 years old (including 18 and 55 years old);
* Male subjects weigh no less than 50 kg. Female subjects weighed no less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), and the body mass index is within the range of 18.0-28.0 (including the cut-off value).

Exclusion Criteria:

* Abnormal conditions judged by clinicians to be clinically significant, which the research doctor considers not suitable for participants;
* A positive test results for hepatitis B virus（HBV）, hepatitis C virus（HCV）, HIV or syphilis;
* Those who have a history of specific allergies or allergies, or those who are known to be allergic to curcumin components or the like;
* A history of alcoholism ;
* A history of dysphagia or any gastrointestinal disease that affects drug absorption;
* Female subjects are breastfeeding during the screening period or clinical trials or have a positive pregnancy test result;
* Those who have a positive drug screening test or have a history of drug abuse in the past five years or have used drugs in the 3 months before taking the drug;
* Those who smoked more than 5 cigarettes a day on average in the 3 months before the test;
* Donate blood or blood loss ≥ 400ml within 3 months before taking the study drug;
* Have a history of surgery or have taken the study drug within 3 months before taking the study drug;
* Any prescription drugs taken within 14 days before taking the study drug;
* Any over-the-counter medicines, herbal medicines or prescribe products taken within 7 days before taking the study drug;
* Have taken a special diet or strenuous exercise or other drugs that affect the study within 48 hours before taking the study drug Those with factors such as absorption, distribution, metabolism, and excretion;
* Consume chocolate, any caffeine-containing or xanthine-rich beverage or food (such as animal liver) within 48 hours before taking the study drug;
* Those who have taken any alcohol-containing products within 24 hours before taking the study medication, or those who have been tested positive for alcohol;
* Subjects judged by other researchers to be unsuitable to participate.

Ages: 18 Years to 55 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Cmax（Peak Plasma Concentration ） | Day 0 to Day 3
  Maximum observed concentration,occurring at Tmax
AUC（AUC0-t，AUC0-∞） | Day 0 to Day 3
  Area under the plasma concentration versus time curve
Tmax | Day 0 to Day 3
  Time of Cmax
F | Day 0 to Day 3
  The rate and extent at which a drug is absorbed into the circulation of the body

SECONDARY OUTCOMES:
tl/2 | Day 0 to Day 3
  Terminal half-life
λz | Day 0 to Day 3
  First Order Terminal Elimination Rate Constant

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Master, Study Director — Qingdao University Hospital
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shangdong, China

IPD SHARING:
Plan to Share IPD: No